CLINICAL TRIAL: NCT02940600
Title: Pilot, Open, Monocentric, Randomized, Prospective Trial for the Evaluation of the Efficacy of Normothermic Perfusion Machine for Organ Preservation in Liver Transplantation Using Brain Death Donors Older or Equal Than 70 Years
Brief Title: Efficacy Evaluation of Normothermic Perfusion Machine Preservation in Liver Transplant Using Very Old Donors
Acronym: CEFEMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Davide Ghinolfi, Medical Doctor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 687
Record Dates: First submitted 2016-10-16; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Reperfusion Injury
Keywords: normothermic perfusion; old donors; extended criteria grafts; reconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normothermic machine perfusion (Experimental): Patients undergoing liver transplant with grafts preserved using normothermic machine perfusion
  Interventions: Device: Normothermic machine perfusion
- Static cold storage (Active Comparator): Patients undergoing liver transplant with statically cold preserved grafts
  Interventions: Procedure: Static cold storage

INTERVENTIONS:
Device: Normothermic machine perfusion — Patients undergoing liver transplant with the use of grafts preserved with normothermic perfusion machine
  Other Names: Liver Assist
  Arms: Normothermic machine perfusion
Procedure: Static cold storage — Patients undergoing liver transplant using statically cold preserved grafts
  Arms: Static cold storage

SUMMARY:
The purpose of this study is to evaluate the impact of normothermic machine perfusion in liver transplantation using grafts of brain death donors older or equal than 70 years

DETAILED DESCRIPTION:
Mean donor age for liver transplantation in Tuscany, Italy, is increasing and is actually 71 years. Old donors are a valuable resource but their use has been related to a major incidence of primary non function (PNF), delayed graft function (DGF) and ischemic type biliary lesions (ITBL).

Ischemia-reperfusion injury is a major reason for the development of these complications and and old grafts are more susceptible than younger ones.

Normothermic machine perfusion (NMP) is a novel and promising technique that allows preservation in a more physiological environment. It is our belief that the use of NMP might reduce the impact of ischemia-reperfusion injuries in older grafts thus reducing the incidence of complications and providing a better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient on waiting list for liver transplant
* Signed informed consent
* Age between 18 and 70
* Eligibility for liver transplant as for University of Pisa Liver Transplant Center Protocol
* Capacity and willingness to participate to the protocol

Exclusion Criteria:

* No signed informed consent
* Age under 18 or over 70
* Presence of disease that may influence results
* Patient participation to other studies
* Re-liver transplant
* ABO incompatible OLT
* Multiorgan transplant
* Liver transplant for acute liver failure or trauma
* MELD (model for end stage liver disease) >24
* Patient not suitable to participate on investigators's opinion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
6 months graft survival | 180 days

SECONDARY OUTCOMES:
Ischemia-reperfusion injury assessment through biopsies evaluation | 1 day
ischemia reperfusion injury assessment through transaminases | 7 days
  AST level at post operative day number 7
Ischemia reperfusion injury assessment through incidence of ischemic type biliary lesions | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Davide Ghinolfi, MD, PhD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- UO Chirurgia Epatica e del Trapianto di Fegato, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bral M, Gala-Lopez B, Bigam D, Kneteman N, Malcolm A, Livingstone S, Andres A, Emamaullee J, Russell L, Coussios C, West LJ, Friend PJ, Shapiro AM. Preliminary Single-Center Canadian Experience of Human Normothermic Ex Vivo Liver Perfusion: Results of a Clinical Trial. Am J Transplant. 2017 Apr;17(4):1071-1080. doi: 10.1111/ajt.14049. Epub 2016 Dec 9. PMID 27639262
- [Background] Mergental H, Perera MT, Laing RW, Muiesan P, Isaac JR, Smith A, Stephenson BT, Cilliers H, Neil DA, Hubscher SG, Afford SC, Mirza DF. Transplantation of Declined Liver Allografts Following Normothermic Ex-Situ Evaluation. Am J Transplant. 2016 Nov;16(11):3235-3245. doi: 10.1111/ajt.13875. Epub 2016 Jul 13. PMID 27192971
- [Background] Op den Dries S, Karimian N, Westerkamp AC, Sutton ME, Kuipers M, Wiersema-Buist J, Ottens PJ, Kuipers J, Giepmans BN, Leuvenink HG, Lisman T, Porte RJ. Normothermic machine perfusion reduces bile duct injury and improves biliary epithelial function in rat donor livers. Liver Transpl. 2016 Jul;22(7):994-1005. doi: 10.1002/lt.24436. PMID 26946466
- [Background] Ravikumar R, Jassem W, Mergental H, Heaton N, Mirza D, Perera MT, Quaglia A, Holroyd D, Vogel T, Coussios CC, Friend PJ. Liver Transplantation After Ex Vivo Normothermic Machine Preservation: A Phase 1 (First-in-Man) Clinical Trial. Am J Transplant. 2016 Jun;16(6):1779-87. doi: 10.1111/ajt.13708. Epub 2016 Mar 7. PMID 26752191